CLINICAL TRIAL: NCT01831063
Title: Simulation for Family Centered Care: Improving Caregivers Skills, Self-Efficacy and Quality of Life Using a Practice-Until-Perfect Simulation Intervention for Seizure Management in the Home Environment
Brief Title: A Simulation-based Intervention for Caregivers of Children With Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Cheng, Director of Research and Development ASPIRE/KidSIM Simulation Program Alberta Children's Hospital, Associate Professor Pediatrics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Alberta Children's Hospital
Record Dates: First submitted 2013-04-01; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Dependency on Medications Prescribed for Patient; Types of Seizures and Epileptic Syndromes
Keywords: Seizure; Caregivers; Family Centered Care; Learning modality
MeSH Terms: conditions — Epileptic Syndromes; Seizures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): This group received the traditional seizure teaching. This consisted of verbal instruction from health care professionals on acute seizure management and administration of the rescue medication.
- 2 (Experimental): This group received the traditional seizure teaching as well as the supplemental simulation based seizure management teaching. The simulation based seizure teaching consisted of numerous opportunities to manage a simulated seizure with instructor guidance and feedback. This session was deemed complete when caregivers verbalized confidence with seizure management.
  Interventions: Behavioral: Simulation

INTERVENTIONS:
Behavioral: Simulation — The experimental group received a simulation based seizure teaching session in addition to the traditional seizure teaching
  Arms: 2

SUMMARY:
Caregivers of children with seizures receiving simulation based seizure management teaching in addition to the traditional seizure teaching will report more confidence with seizure management and demonstrate a higher level of performance with seizure management.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of Seizure disorder
* Dependence on a anti-seizure medication

Exclusion Criteria

* No dependence on rescue medication

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
KidSIM Emergent Seizure Management Checklist | Baseline, 48 hours and 6 months
  Caregivers performance managing a seizure scenario was assessed at baseline and at 48 hours after which time caregivers received their respective teaching sessions. Caregivers in the both groups participated in the traditional seizure teaching sessions. Caregivers in the intervention group received an additional simulation-based seizure teaching session that consisted of opportunities to practice seizure management in a simulated environment with instructor feedback and guidance. These sessions generally lasted 30 minutes and were deemed complete when caregivers were able to verbalize confidence with seizure management. The performance of caregivers in both groups were assessed again immediately after they received their respective teaching sessions which was usually the day of discharge.

SECONDARY OUTCOMES:
The Aspire KidSIM Parent Seizure Self-efficacy Questionnaire | Baseline , 48 hours and 6 months
  Caregivers were asked to fill out the questionnaire at baseline and after they received their respective teaching sessions which was at 48 hours post baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Sigalet, PhD, Principal Investigator — Alberta Children's Hospital; Vincent Grant, MD, Principal Investigator — Alberta Children's Hospital, University of Calgary; Adam Cheng, MD, Principal Investigator — Alberta Children's Hospital, University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada